CLINICAL TRIAL: NCT06804200
Title: Prospective Validation of AKI Prediction Algorithm
Brief Title: Prospective Validation of AKI Prediction
Status: Not yet recruiting | Type: Observational
Sponsor: Adam C Dziorny (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Adam C Dziorny, Associate Professor of Pediatrics, University of Rochester
Organization: University of Rochester (Other)
Other Study IDs: STUDY00008612; K23DK138299 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Acute Kidney Injury
Keywords: Machine Learning; Pediatrics; Critical Care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric ICU Admissions: The study subjects are all patients admitted to the pediatric intensive care unit and the pediatric cardiac care unit at Golisano Children's Hospital at Strong. By virtue of admission to a pediatric hospital bed, all subjects will be children. The rationale for focusing on this population is that the developed algorithm focuses on identifying acute kidney injury among critically ill pediatric patients. The gender and age of subjects will not influence enrollment. To accurately determine algorithm test characteristics (sensitivity, PPV, NNA) pragmatically, Investigators must include all admitted patients. Missing patients may bias our results and invalidate the study.

SUMMARY:
The purpose of this prospective observational study is to implement, deploy, and quantify accuracy of an existing Pediatric Early AKI Risk Score algorithm. The implementation will be facilitated using a Health Level 7 (HL7) Fast Healthcare Interoperability Resource (FHIR)-based architecture. Investigators will deploy this model and store results in a manner not viewable to the clinical team caring for the patient. To determine the accuracy of the implemented prediction model, Investigators will prospectively identify patients with AKI at 72 hours following ICU admission. Investigators hypothesize that this model will prospectively detect AKI with a sensitivity >70% and a positive predictive value >20%, both chosen a priori as 10% improvement over the initial Pediatric AKI Risk Score tool.

DETAILED DESCRIPTION:
This is a single-center prospective observational study validating an AKI predictive model. Each model feature will be mapped to an appropriate FHIR-based resource. To mitigate the latency issues seen in other distributed CDS systems, Investigators have developed an asynchronous design where algorithm calculations are performed offline (e.g., not within the EHR) and risk scores are subsequently written back to the EHR. Importantly, in this deployment, model output and resulting clinical risk score will not be communicated to the treating clinicians.

During the study period, Investigators will review charts daily for all patients admitted to the Golisano Children's Hospital PICU, a 12-bed facility adjacent to our 15-bed Pediatric Cardiac Intensive Care Unit (PCICU). Using a standard protocol to screen and identify patients by chart review, Investigators will generate a list of patients who meet AKI KDIGO criteria by SCr and urine output, along with recorded clinical information about these patients. At the conclusion of the study period, this list will be used as the "gold standard" and compared to the automated screening tool to determine the tool's test characteristics.

Model assessment outcomes include sensitivity, positive predictive value (PPV), and number needed to alert (NNA) to prospectively identify AKI in a population of critically ill children. Additional outcomes include timeliness of identification based on model implementation (e.g., measured timestamps of algorithm prediction compared to manual, prospectively identified AKI development). Additionally, Investigators will report interventions and clinical outcomes of the prospectively identified patients with AKI, stratified by those predicted early by the model (within 24 hours of admission) versus not.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Pediatric Intensive Care Unit or Pediatric Cardiac Intensive Care Unit
* Age > 30 days and < 18 years

Exclusion Criteria:

* Discharged less than 12 hours after admission
* AKI at 12 hours of admission by KDIGO Serum Criteria

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All medical and surgical patients admitted to the pediatric intensive care unit and pediatric cardiac intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury (AKI) within the first 72 hours of ICU admission | Within 72 hours following ICU Admission
  Acute Kidney Injury (AKI) defined by KDIGO stages 1, 2, or 3, based on changes in serum creatinine levels or urine output (UOP), assessed within the first 72 hours of ICU admission. Stage 1 is defined by a 1.5 to 1.9 times baseline serum creatinine or an increase of ≥0.3 mg/dL. Stage 2 is a 2.0 to 2.9 times baseline increase, and Stage 3 is a 3.0 times baseline increase or a serum creatinine ≥4.0 mg/dL.

SECONDARY OUTCOMES:
Prediction Accuracy and Timeliness of AKI Risk using a Predictive Model | Within 12 hours of ICU Admission
  Predictive model results generated prospectively (at 12 hours following admission) will be used to generate a 2x2 confusion matrix with prospectively identified AKI by serum creatinine or urine output changes based on KDIGO criteria. Investigators will calculate sensitivity, PPV, and NNA for the prospective identification of AKI. Investigators will report the time of AKI prediction compared to admission date and the onset date of AKI.
Risk of Mortality in Patients with Acute Kidney Injury (AKI) | 28 Days following ICU admission
  Investigators will assess for AKI independent risk of mortality at 28 days after adjusting for confounders.

CONTACTS AND LOCATIONS:
Locations (1):
- Golisano Children's Hospital at Strong, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Non-PHI data elements may be made available by request, per data sharing plan.